CLINICAL TRIAL: NCT05081648
Title: A Randomised Control Trial of MuST Technique for Vascular Access Cannulation in Hemodialysis Patients: Contributions for a Safe Nursing Intervention
Brief Title: Must Cannulation Technique of Vascular Access in Patients Undergoing Haemodialysis: Contributions for a Safe Nursing Intervention
Acronym: MuST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: University of Lisbon (Other); Lisbon School of Nursing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD-MuST-01-PT
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Diseases; Hemodialysis; Vascular Access Complication; Hemodialysis Access Failure; Arteriovenous Fistula
Keywords: Chronic Kidney Disease; Hemodialysis; Vascular access; Vascular Access Complication; Rope-ladder; Cannulation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: multiple-center, prospective, non-blind, parallel-group, randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Multiple Single Cannulation Technique (MuST) (Experimental)
  Interventions: Procedure: CT MuST
- Control group: Rope-ladder cannulation technique (RL) (Other)
  Interventions: Procedure: Rope-ladder cannulation technique

INTERVENTIONS:
Procedure: CT MuST — Multiple Single Cannulation Technique (MuST): Experimental technique
  Arms: Intervention group: Multiple Single Cannulation Technique (MuST)
Procedure: Rope-ladder cannulation technique — Standard cannulation technique( Rope-ladder)
  Arms: Control group: Rope-ladder cannulation technique (RL)

SUMMARY:
The aims of this study are to:

* Determine the AVF (arteriovenous fistula) survival of patients submitted to MuST compared to those submitted to RL (rope-ladder).
* Determine the AVF (arteriovenous fistula) complication rate of patients submitted to MuST compared to those submitted to RL (rope-ladder).
* Analyze the intensity of pain perceived by the patient with each cannulation technique under study.

DETAILED DESCRIPTION:
The MuST is based on the association between the RL technique in that it uses the entire length of the available vessel through progressive rotation, and the buttonhole (BH) cannulation technique since there are three specific cannulation sites for each cannulation day during the week, meaning that each site is only cannulated once a week (allowing the puncture site to heal in between cannulations).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the study and sign an informed consent;
* Are on a regular haemodialysis (HD) program with three weekly sessions;
* AVF has been in use for at least 4 weeks without incident;
* AVF with blood flow (Qa) ≥500 mL/min evaluated by thermodilution;
* AVF paths allow cannulations along the entire length of the vein with at least 6 cm of distance between bevels, or two distinct areas of 3 cm in length;
* Adult patients

Exclusion Criteria:

* Those who decline to take part;
* Those who have undergone angiography or surgical intervention in the last 4 months in the AVF in use;
* Those who have undergone three or more interventions in the AVF in use;
* Those with use of anesthetic creams at cannulation sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Vascular access survival rate | 12 months after start of study
  Vascular access (VA) survival rate at 12 months and determined by the percentage of fistulas in use from the beginning of the study to the date of the first clinical intervention by angioplasty or vascular surgery, to maintain or restore patency - "unassisted patency".

SECONDARY OUTCOMES:
Arteriovenous fistula survival rate | 12 months after start of study
  Arteriovenous fistula (AVF) survival rate at 12-month and determined by the percentage of fistulas in use from the study start to the date of access abandonment due to dysfunction, patient abandonment, or death, treatment change modality or study end.

CONTACTS AND LOCATIONS:
Locations (3):
- Portugal (3):
  - NephroCare Coimbra, Coimbra
  - Nephrocare Montijo, Montijo
  - NephroCare Vila Nova de Gaia, Vila Nova de Gaia

REFERENCES:
- [Derived] Peralta R, Wammi A, Stauss-Gabo M, Dias O, Carvalho H, Cristovao A. A randomised control trial protocol of MuST for vascular access cannulation in hemodialysis patients (MuST Study): contributions for a safe nursing intervention. BMC Nephrol. 2022 Jun 21;23(1):218. doi: 10.1186/s12882-022-02842-3. PMID 35729492